CLINICAL TRIAL: NCT05906979
Title: Digital Human-Based Brief Interventions for Harmful Alcohol Use: The PAHOLA Project
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Pan American Health Organization (Other)
Responsible Party: Principal Investigator, Jurgen Rehm, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-0615
Record Dates: First submitted 2023-05-29; First posted 2023-06-18 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Alcohol Drinking; Alcoholism
MeSH Terms: conditions — Alcohol Drinking; Alcoholism | interventions — Ethanol; Health

STUDY DESIGN:
Intervention Model Description: a pilot RCT will be performed where the first group will receive a BI, the second group will receive a text-only version of PAHO's BI, and the third group will receive information from PAHOLA about the risks of alcohol use.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Digital intervention (Experimental): Participants will interact with PAHOLA the digital assistant of the Pan American Health Organization.
  Interventions: Other: PAHOLA (digital health assistant)
- Digital intervention (text only) (Experimental): Participants will interact with PAHOLA (text only version) the digital assistant of the Pan American Health Organization.
  Interventions: Other: PAHOLA (digital health assistant)
- Information on alcohol use and risk (Other): A PDF containing standard information on alcohol use and risk from the Pan American Health Organization.
  Interventions: Other: Standard information on alcohol use and health

INTERVENTIONS:
Other: PAHOLA (digital health assistant) — Pahola is the Pan American Health Organization's new digital health specialist on alcohol use. Programmed with the latest information and research, she can help you make healthier decisions related to your alcohol consumption. Pahola is free to use and can easily be accessed from the privacy of your own home by making use of the online app.
  Arms: Digital intervention; Digital intervention (text only)
Other: Standard information on alcohol use and health — A brochure on alcohol use and health as produced by the Pan American Health Organization will be provided to participants.
  Arms: Information on alcohol use and risk

SUMMARY:
Alcohol use disorders are among the most prevalent mental disorders in Canada; however, due to numerous barriers, including fear of treatment, privacy concerns, stigma, time conflicts, and lack of availability of treatment, less than 10% of people with alcohol dependence receive treatment. Accordingly, there is a need to expand treatment coverage for alcohol use disorders, especially for populations which face barriers to receiving treatment.

The objective of this proposed project is to develop a digital health worker, named PAHOLA, which can effectively deliver interventions to people who would not otherwise receive such treatment. To achieve this objective, the following research aims will be addressed:

1. To develop a digital human-based intervention that can initiate change processes and reduce alcohol use by applying the principles of motivational interviewing (MI) and cognitive behavioural therapy (CBT) in a credible manner.
2. To assess the impact of the virtual care provided by PAHOLA on health outcomes using a randomized controlled study design (RCT) to assess potential effect sizes for a larger future RCT.

If successful, the PAHOLA project has the potential to transform our ability to prevent alcohol-attributable harms in Canada by promoting health, health equity, and well-being, especially among those people who do not normally receive treatment for harmful alcohol use.

DETAILED DESCRIPTION:
Alcohol use disorders are among the most prevalent mental disorders in Canada; however, due to numerous barriers, including fear of treatment, privacy concerns, stigma, time conflicts, and lack of availability of treatment, less than 10% of people with alcohol dependence receive treatment. Accordingly, there is a need to expand treatment coverage for alcohol use disorders, especially for populations which face barriers to receiving treatment.

.

The objective of this proposed project is to tailor PAHOLA into a digital health worker which can effectively deliver BIs to people who would not otherwise receive such treatment. To achieve this objective, the following research aims will be addressed:

3. To develop a digital human-based intervention that can initiate change processes and reduce alcohol use by applying the principles of motivational interviewing (MI) and cognitive behavioural therapy (CBT) in a credible manner.

4. To assess the impact of the virtual care provided by PAHOLA on health outcomes using a randomized controlled study design (RCT) to assess potential effect sizes for a larger future RCT.

To address these objectives, the study will employ the following research strategy

This project will build upon the PAHOLA digital human prototype which was developed by Soul Machines, the Pan American Health Organization (PAHO), and Rooftop to provide information on alcohol risks and harms. This project will develop PAHOLA to intervene in cases of hazardous and harmful alcohol use, and will take place in the following three phases:

Phase 1 - development of the intervention dialogue flow program. PAHOLA will (i) screen for harmful alcohol use using the AUDIT, and (ii) deliver Brief Intervention (BIs). The BIs will be based primarily on two evidence-based approaches that are used to effectively treat alcohol misuse, namely MI and CBT. Dialogue will be constructed in alignment with FRAMES - Feedback, Responsibility, Advice, Menu of options, Empathy, and Self efficacy (confidence for change),and OARS - (Open ended questions, Affirmation, Reflective listening, and Summarizing).

Phase 2 - a two-day virtual meeting of researchers, health care providers, and people with lived experience. A virtual meeting of a total of 30 experts will be held to comment upon and further develop PAHOLA. Meeting participants will formulate a series of evidence-based recommendations regarding how to improve: 1) the affinity and trustworthiness of PAHOLA, 2) the dialogue flow for BIs, and 3) the specific dialogue flows for men and women.

Phase 3 - a pilot randomized controlled trial (RCT) of the PAHOLA intervention program. To assess PAHOLA as a potential intervention for treating harmful alcohol use, a pilot RCT will be performed where the first group will receive a BI, the second group will receive a text-only version of PAHO's BI, and the third group will receive information from PAHOLA about the risks of alcohol use. A total of 180 adults (18 years of age and older) with hazardous and harmful alcohol use will be recruited via online advertisements and databases of individuals interested in participating in research studies.

ELIGIBILITY:
Inclusion Criteria:

1. Current drinkers 18 years of age and older who score 7 to 23 on the Alcohol Use Disorders Identification Test
2. Use of medication to treat harmful alcohol use will be allowed provided that the dose has been stable for 8 weeks
3. Availability of a computer with a connection to the internet and a camera and microphone

Exclusion Criteria:

1. A history of drug use disorders (other than alcohol) in the last two years (except tobacco use disorder)
2. Dose changes of concomitant medications will not be permitted during the study period
3. Pregnant or lactating women, and women of childbearing potential who are not using medically accepted forms of contraception, or women who are planning on becoming pregnant during the study time frame
4. People who are currently reciving psychological treatment for alcohol use disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes in alcohol use quantity | 1 month
  Alcohol use quantity (measured in average grams per day in the past week)
Changes in alcohol use quantity | 3 months
  Alcohol use quantity (measured in average grams per day in the past week)
Changes in alcohol use quantity | 6 months
  Alcohol use quantity (measured in average grams per day in the past week)
Changes in alcohol use frequency | 1 month
  Alcohol use frequency (measured in drinking days in the past week)
Changes in alcohol use frequency | 3 months
  Alcohol use frequency (measured in drinking days in the past week)
Changes in alcohol use frequency | 6 months
  Alcohol use frequency (measured in drinking days in the past week)
Changes in Alcohol Use Disorders Identification Test (AUDIT) items 5 to 10 scores | 1 month
  Alcohol Use Disorders Identification Test (AUDIT) items 5 to 10 scores; Scale (0 to 15); Higher scores indicate harmful alcohol use.
Changes in Alcohol Use Disorders Identification Test (AUDIT) items 5 to 10 scores | 3 months
  Alcohol Use Disorders Identification Test (AUDIT) items 5 to 10 scores; Scale (0 to 15); Higher scores indicate harmful alcohol use.
Changes in Alcohol Use Disorders Identification Test (AUDIT) items 5 to 10 scores | 6 months
  Alcohol Use Disorders Identification Test (AUDIT) items 5 to 10 scores; Scale (0 to 15); Higher scores indicate harmful alcohol use.

SECONDARY OUTCOMES:
Changes in anxiety | 1 months
  Hamilton Anxiety Rating Scale (HAM-A) 36; Scale range: 0-56; Higher scores indicate worse anxiety
Changes in anxiety | 3 months
  Hamilton Anxiety Rating Scale (HAM-A) 36; Scale range: 0-56; Higher scores indicate worse anxiety
Changes in anxiety | 6 months
  Hamilton Anxiety Rating Scale (HAM-A) 36; Scale range: 0-56; Higher scores indicate worse anxiety
Changes in depression | 1 months
  Patient Depression Questionnaire - 9 item version; Scale range: 0 to 27; Higher scores indicate worse depression
Changes in depression | 3 months
  Patient Depression Questionnaire - 9 item version; Scale range: 0 to 27; Higher scores indicate worse depression
Changes in depression | 6 months
  Patient Depression Questionnaire - 9 item version; Scale range: 0 to 27; Higher scores indicate worse depression
Changes in quality of life | 1 month
  Short Form Health Survey-12 item (SF-12); Scale range: 0 to 100; Higher scores indicating better physical and mental health functioning.
Changes in quality of life | 3 months
  Short Form Health Survey-12 item (SF-12); Scale range: 0 to 100; Higher scores indicating better physical and mental health functioning.
Changes in quality of life | 6 months
  Short Form Health Survey-12 item (SF-12); Scale range: 0 to 100; Higher scores indicating better physical and mental health functioning.
Packs of cigarettes smoked in the past week | 1 month
  Packs of cigarettes smoked in the past week
Packs of cigarettes smoked in the past week | 3 months
  Packs of cigarettes smoked in the past week
Packs of cigarettes smoked in the past week | 6 months
  Packs of cigarettes smoked in the past week

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Shield, Principal Investigator — Centre for Addiction and Mental Health

IPD SHARING:
Plan to Share IPD: No